CLINICAL TRIAL: NCT05876533
Title: An Observational, Retrospective, Single-arm, Open US and Israel Study , for Usability Assessment and Algorithm, Development of the Cordio HearO™ Systeam
Brief Title: R&D Study to Evaluate Cordio's Usability and to Collect Patient Speech Utterances
Status: Active, not recruiting | Type: Observational
Sponsor: Cordio Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: CLN0016
Record Dates: First submitted 2023-04-23; First posted 2023-05-25 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Chronic Heart Failure
Keywords: CHF

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Device: Cordio HearO — Cordio HearO is a software medical device that remotely monitors Congestive Heart Failure (CHF) patients by detecting changes in the patients' recorded voice relative to a baseline. The system is comprised of a mobile application (or "app") that is deployed on a mobile platform, and a web-based portal that enables caregivers to manage their patients

SUMMARY:
To determine the usability and technical aspects of Cordio HearO™

DETAILED DESCRIPTION:
The system (including App and server) will be tested under simulated use conditions with representative users to identify potential changes required to the application user interface, to improve user performance and satisfaction, and to inform future design options.

The recordings data will also be used for algorithm improvement

ELIGIBILITY:
Major inclusion Criteria:

1. Adults patients
2. Diagnosed with Symptomatic Chronic Heart Failure [NYHA II-IVa (ambulatory)]
3. At least one of the following:

   1. One ADHF hospitalization in the last 12 months
   2. One unplanned IV/SC diuretic administration in the last 6 months
   3. Two unplanned IV/SC diuretic administration in the last 12 months
   4. NTProBNP >500 pg/ml or BNP*> 150 pg/ml at screening visit
4. Clinically stable HF
5. Willing to participate as evidenced by signing the written informed consent.
6. Male or non-pregnant female patient (pre-menopausal women will confirm verbally).

Major exclusion Criteria:

1. Not able to read in Hebrew, Russian, Arabic, English and/or Spanish.
2. Unable to comply with daily use of the App
3. Major cardiovascular event
4. Had a Cardiac Resynchronization Device (CRT) implanted or upgrading ≤ 1 month prior to screening visit.
5. Has estimated Glomerular Filtration Rate (eGFR) < 30 ml/min/1.73 meter square (Cockroft-Gault formula).
6. Is likely to undergo heart transplantation/ LVAD within 6 months of Screening Visit.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult clinical stable patients with NYHA II-IVa (ambulatory)
Sampling Method: Non-Probability Sample
Enrollment: 216 (Actual)
Dates: Start 2022-03-18 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-03-15 (Estimated)

PRIMARY OUTCOMES:
Patient Usability success defined as: 1.Total and individual usability score of ≥3 in the usability questionnaire in ≥80% of the users. | 2 years
  The used scale is: Usability questionnaire for the Cordio HearO™ App. This Usability questionnaire is a subjective evaluation based on Likert score of device user satisfaction.
  Maximum value for each item: 5 Minimum value for each item: 1 Higher scores means a better outcome
Patient Usability success defined as: 2. Total Compliance | 2 Years
  The total compliance will be determined by the total number of recording days. Success will be considered if total average compliance of 70 % of all days.

CONTACTS AND LOCATIONS:
Overall Officials: Ronit Haviv, PhD, Study Director — Cordio Medical
Locations (7):
- United States (4):
  - Kurker Family Medicine, South Windsor, Connecticut
  - C&R Research Services, Cape Coral, Florida
  - C&R Research Services, Miami, Florida
  - Lake County Med Grp, Athens, Georgia
- Israel (3):
  - Barzilai Medical Center- Cardiology, Ashkelon
  - Heart Failure Clinic - Clallit Be'er Sheva, Beersheba
  - Rabin Medical Center - Cardiology- CHF, Petah Tikva